CLINICAL TRIAL: NCT03822338
Title: Pneumoperitoneum Preconditioning for the Prevention of Renal Function After Laparoscopic Partial Nephrectomy: a Double-blind Randomized Controlled Trial
Brief Title: Pneumoperitoneum Preconditioning for the Prevention of Renal Function After Laparoscopic Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ruipeng Jia, Study Chair, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NFH20180205
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Ischemia Reperfusion Injury
Keywords: Renal ischemia reperfusion injury; Pneumoperitoneum preconditioning; Laparoscopic partial nephrectomy
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumoperitoneum preconditioning group (Experimental): Participant assigned to the this group will receive a treatment consisting of three cycles of 5 min insufflation (intra-abdominal pressure at 15 mmHg) and 5 min desufflation, after complete anesthesia and successfully implanting the veress.
  Interventions: Procedure: Pneumoperitoneum preconditioning
- Control group (Sham Comparator): Participants in the control group will receive the same placement of the veress but without insufﬂation and subsequent desufﬂation.
  Interventions: Procedure: Sham-Pneumoperitoneum preconditioning

INTERVENTIONS:
Procedure: Pneumoperitoneum preconditioning — Pneumoperitoneum preconditioning consists of three cycles of 5 min insufflation and 5 min desufflation, after complete anesthesia and successfully implanting the veress. This process will be induced by pneumoperitoneum machine, and the utilized gas will be carbon dioxide to maintain the intra-abdominal pressure at 15 mmHg. The whole duration will last 30 min.
  Arms: Pneumoperitoneum preconditioning group
Procedure: Sham-Pneumoperitoneum preconditioning — Sham-Pneumoperitoneum preconditioning consists of three cycles without insufﬂation and subsequent desufﬂation. The whole duration will also last 30 min.
  Arms: Control group

SUMMARY:
The present study is designed to investigate the short-term and long-term renoprotective role of pneumoperitoneum preconditioning in patients undergoing laparoscopic partial nephrectomy.

DETAILED DESCRIPTION:
Renal ischemia reperfusion injury (IRI) is an inevitable event in patients undergoing laparoscopic partial nephrectomy (LPN), which can obviously affect the post-operational renal function. Pneumoperitoneum preconditioning (PP) is a promising strategy to render a protective effect on kidney, which has been already confirmed in some clinical settings. This study is designed as a randomized, prospective, double-blind and parallel controlled clinical trial to assess the short-term and long-term renoprotective role of pneumoperitoneum preconditioning in patients undergoing laparoscopic partial nephrectomy, and observe its effect on the other abdominal organs. Patients with renal tunours and willing to accept elective LPN will be screened as eligible participants. The investigators aim to enroll 86 subjects. Patients randomized to the treatment arm will receive PP consisted of three cycles of 5 min insufﬂation and 5 min desufﬂation before PLN, while the control arm receive a sham operation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older;
* Patients with renal tumours (whether benign or malignant) and accept laparoscopic partial nephrectomy as the surgical method;
* The renal tumor must be stage T1a (assessed by MRI/CT), and tumor≤4cm in diameter;
* Unilateral renal tumour, and another contralateral renal function reveal normal (renal function >40% as determined by radionuclide scintigraphy);
* Patients volunteer for this study and provided written informed consent.

Exclusion Criteria:

* Large tumour (tumor>4cm in diameter);
* Severe renal insufficiency (glomerular filtration rate, GFR<30 ml/min/1.73m2) or needing preoperative dialysis (hemodialysis or peritoneal dialysis);
* Patients severe cardiopulmonary dysfunction;
* Pregnancy Women;
* Patients with other malignant tumours;
* Patients who have had a renal transplantation;
* Patients with a history of other abdominal viscera operations within one year (open or under laparoscope);
* American Society of Anesthesiologists (ASA)>Ⅲ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The absolute change in glomerular filtration rate (GFR) | changes from baseline and postoperative 1, 6 months
  Unilateral and overall GFR detected by 99mTc-DTPA renal scintigraphy.
The absolute change in the level of serum Cystatin C (Cys C) | changes from baseline and 12, 24, 48 hours after desufflation
  The absolute change in the level of serum Cys C after desufflation.

SECONDARY OUTCOMES:
The level of serum creatinine (SCr) | Baseline; 12, 24, 48 hours, and 1, 6 months after desufflation
  The absolute change in the level of serum SCr after desufflation.
Estimated glomerular filtration rate (eGFR) | Baseline; 12, 24, 48 hours, and 1, 6 months after desufflation
  eGFR will be calculated by a combined formula.
The level of alanine transaminase (ALT) | Baseline; 12, 24, 48 hours, and 1, 6 months after desufflation
  Serum markers for detecting the insults of the liver.
The level of serum amylase | Baseline; 12, 24, 48 hours, and 1, 6 months after desufflation
  Serum markers for detecting the insults of the pancreas.
The level of intestinal fatty acid binding protein (I-FABP) | Baseline; 12, 24, 48 hours, and 1, 6 months after desufflation
  Serum markers for detecting the insults of the intestine.

OTHER OUTCOMES:
Duration of postoperative hospital stay | 6 months following surgery
Incidence of adverse events | 6 months following surgery
Rate of mortality | 6 months following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou C, Xu L, Xu Z, Ge Y, Zhou L, Wang F, Liu J, Pan G, Yang T, Jia R. Pneumoperitoneum preconditioning for the prevention of renal function after laparoscopic partial nephrectomy: protocol for a double-blind randomised controlled trial. BMJ Open. 2020 May 26;10(5):e032002. doi: 10.1136/bmjopen-2019-032002. PMID 32461289